CLINICAL TRIAL: NCT04289064
Title: Artificial Intelligence System for Assessing Image Quality of Fundus Images and Its Effects on Diagnosis: A Clinical Trial
Brief Title: Artificial Intelligence System for Assessing Image Quality of Fundus Images and Its Effects on Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Other Study IDs: IMAQUA2020-China-01
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Retinal Diseases; Artificial Intelligence
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fundus image quality assessment: Device: an artificial intelligence system for quality assessment of fundus images. These patients are enrolled in primary healthcare units or the AI clinic at Zhongshan Ophthalmic Center.
  Interventions: Device: Taking a fundus image

INTERVENTIONS:
Device: Taking a fundus image — The participant only needs to take a fundus image as usual.

SUMMARY:
Fundus images are widely used in ophthalmology for the detection of diabetic retinopathy, glaucoma and other diseases. In real-world practice, the quality of fundus images can be unacceptable, which can undermine diagnostic accuracy and efficiency. Here, the researchers established and validated an artificial intelligence system to achieve automatic quality assessment of fundus images upon capture. This system can also provide guidance to photographers according to the reasons for low quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be aware of the contents and signed for the informed consent.

Exclusion Criteria:

* 1. Patients who cannot cooperate with a photographer such as some paralytics, the patients with dementia and severe psychopaths.
* 2. Patients who do not agree to sign informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria:
  * Patients should be aware of the contents and signed for the informed consent.
  Exclusion Criteria:
  * 1. Patients who cannot cooperate with a photographer such as some paralytics, the patients with dementia and severe psychopaths.
  * 2. Patients who do not agree to sign informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Performance of artificial intelligence system for distinguish between good image quality and poor image quality | 3 months
  Area under the receiver operating characteristic curves, sensitivity, specificity, positive and negative predictive values, accuracy

SECONDARY OUTCOMES:
The comparison of the performance for previous artificial intelligence diagnostic system with fundus images of different image quality | 3 months
  Cohen's kappa coefficient, P value and other related statistic results

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No